CLINICAL TRIAL: NCT05985837
Title: Post Market Clinical Follow-Up Study on Medical Devices KalobaGola Useful for Sore Throat and/or Pharyngitis in Adults and Children
Brief Title: Post Market Clinical Follow-Up Study - Medical Device KalobaGOLA ( PMCF )
Acronym: PMCF
Status: Completed | Type: Observational
Sponsor: Schwabe Pharma Italia (Industry)
Responsible Party: Sponsor
Other Study IDs: KG-01-2023
Record Dates: First submitted 2023-08-02; First posted 2023-08-14 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Sore-throat; Pharyngitis
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Adolescents and adults: Adolescents from 12 years old and adults with sore throat and/or pharyngitis, who have bought the product.
  Interventions: Device: KalobaGOLA spray (1); Device: KalobaGOLA tablets
- Children 1-6 years: Children from 1 to 6 years old with sore throat and/or pharyngitis, whose parents/caregivers have bought the product.
  Interventions: Device: KalobaGOLA spray (2)
- Children 6-12 years: Children from 6 to 12 years old with sore throat and/or pharyngitis, whose parents/caregivers have bought the product.
  Interventions: Device: KalobaGOLA spray (1); Device: KalobaGOLA tablets

INTERVENTIONS:
Device: KalobaGOLA spray (1) — Oral spray, 2-4 spray, till 8 times per day
  Groups: Adolescents and adults; Children 6-12 years
Device: KalobaGOLA spray (2) — Oral spray, 2-4 spray, till 4 times per day
  Groups: Children 1-6 years
Device: KalobaGOLA tablets — 1 tablets, 6 times per day
  Groups: Adolescents and adults; Children 6-12 years

SUMMARY:
The goal of this observational PMCF study is to confirm the efficacy and safety of the medical device KalobaGola (oral spray and tablets) in children, adolescents and adults with sore throat and /or pharyngitis. The main questions it aims to answer are:

* Is the product effective in the treatment of sore throat / pharyingits?
* Is the product safe?

After buying the product, participants will be asked to fill in a questionnaire, in order to:

1. Assess the sore throat symptoms before the use of the spray or tablets.
2. Assess the resolution of sore throat / pharyngitis symptoms after the use of the spray or tablets.
3. Describe the adverse effect(s)/problem(s) observed while using the product (if any).

DETAILED DESCRIPTION:
The Medical Device Regulation (EU) 2017/745 (MDR) considers post-market clinical follow-up (PMCF) as a continuous process that aims to update the clinical evaluation and validate or reassess the benefit-risk balance of the medical device. The PMCF is an integral part of the manufacturer's post-market surveillance plan (PMS).

The medical devices in question are both CE marked since 2020, with no substantial modification.

The objectives of this Post Market Clinical Follow Up (PMCF) study are: verify the use of these devices in a real situation, verify if their efficacy and safety of use are aligned with the provisions of the clinical evaluation; confirm or reassess the benefit/risk balance; update the risk analysis; identify any need for CAPA.

Specific product questionnaires have been developed based on the validated STAT-10 questionnaire, which aim to investigate aspects of Real-World Evidence on efficacy, safety, even in specific categories or situations, known and unknown adverse events, difficulties in use or completeness and clarity of IFUs.

Given the low-risk class of the devices (class IIa - Dir. 93/42/EEC), which are intended for use by lay people and normally sold in pharmacies / parapharmacies, the sponsor planned to distribute the questionnaires to users that have purchased the product through health professionals (pharmacists), who are normally in charge of the distribution of the products.

The questionnaire was prepared in simple and easily understandable language for lay people.

The data requested during the filling of the questionnaire does not provide for the collection of information that allows the sponsor an identification of the participant.

Data will be collected and processed in a totally anonymous form.

ELIGIBILITY:
Inclusion Criteria:

* KalobaGOLA spray: children from 1 year, adolescents and adults, both sexes, with symptoms of sore throat (burning sensation, pharyngitis, pain on swallowing), who / whose parents or caregivers bought the product by the pharmacy/parapharmacy involved.
* KalobaGOLA tablets: children from 6 years, adolescents and adults, both sexes, with symptoms of sore throat (burning sensation, pharyngitis, pain on swallowing), who / whose parents or caregivers bought the product by the pharmacy/parapharmacy involved.

Exclusion Criteria:

* KalobaGOLA spray: children aged < 1 year, people without sore throat symptoms
* KalobaGOLA tablets: children aged < 6 years, people without sore throat symptoms

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Customers of the pharmacies/parapharmacies involved
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2023-08-02 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Resolution of the symptoms of sore throat / pharyngitis | Before use and at the resolution (after maximum 7 days)
  A 7-items close question questionnaire developed based on STAT-10 (Sore Throat Assessment Tool-10), a validated and published questionnaire. It is a five-points scale with values from 1 to 5 (1= not at all; 5 = very high degree).

SECONDARY OUTCOMES:
Rate of known and unknown side-effects and / or other risks associated to the use of medical devices | During and after use (from the first application to after maximum 7 days)
  Safety of the devices during and after use

CONTACTS AND LOCATIONS:
Locations (1):
- Schwabe Pharma Italia, Neumarkt, Bolzano, Italy